CLINICAL TRIAL: NCT03618745
Title: Outcome Predictors of Non Traumatic Coma in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanan Zaka Saied, Principal investigator, Assiut University
Other Study IDs: Non Traumatic Coma in Children
Record Dates: First submitted 2018-07-20; First posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Impaired Consciousness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CT brain — noninvasive medical examination or procedure that uses specialized X-ray equipment to produce cross-sectional images of the body.

SUMMARY:
To catch the high risk comatosed child to improve service and direct the limited resources to those children in countries with limited resources .

DETAILED DESCRIPTION:
Non Traumatic Coma in children is an important pediatric emergency. It has been an enigma for clinicians for many years. To find the cause of coma and to determine the prognosis is a taxing question for the attending clinicians and the primary concern for relatives in every case.

Non-traumatic coma in childhood accounts for high morbidity and mortality in pediatric age group. It can result from wide range of primary etiologies. Etiology of coma and clinical status at the time of admission are likely outcome predictors. Infection is the commonest etiology for coma in all age groups .

Coma in children is recognized to be a non-specific sign with a wide potential differential diagnosis. Among various etiological factors identified for non-traumatic coma, considerable regional diversity exists in them with infectious problems suggested to be more common in developing countries. There has been few case series in developing countries with specific reference to infective etiology and there are also differences in infective agents between developing and developed countries. Similarly prediction of outcome of coma is difficult early in the course of the illness, especially in children. There have been many studies suggesting prognostic parameters of coma in adults, but limited reviews are available for children.

Etiologically it can be divided into two broad categories: those without focal neurologic signs (e.g., metabolic encephalopathies); meningitis syndromes, characterized by fever or stiff neck and an excess of cells in the spinal fluid (e.g., bacterial meningitis, subarachnoid hemorrhage); and conditions associated with prominent focal signs (e.g., stroke, cerebral hemorrhage). In most instances coma is part of an obvious medical problem such as drug ingestion, hypoxia, stroke, trauma, or liver or kidney failure. Conditions that cause sudden coma include drug ingestion, cerebral hemorrhage, trauma, cardiac arrest, epilepsy, or basilar artery embolism. Coma that appears subacutely is usually related to a preceding medical or neurologic problem, including the secondary brain swelling of a mass lesion such as tumor or cerebral infarction.

Central nervous infections are the most common cause . Toxic-metabolic, status-epilepticus, hypoxic-ischemic, intracranial bleed etc. are other main causes.

Neurological outcome is often the foremost concern of parents and physicians .Etiology of coma and clinical status at the time of presentation are the most likely predictors of outcome. Simple clinical signs have been found as good predictors of outcome .

Non-traumatic coma is an important source of morbidity and mortality in the pediatric age group. Accurate diagnosis of etiology of childhood coma in resource poor countries is complicated by overlap in clinical presentation, limited diagnostic resources, disease endemicity and co-morbidity . Considerable skill is required to distinguish the group at high risk for further deterioration, potentially leading either to death or severe handicap. This study attempts to identify the common etiological factors of pediatric comatose patients as well as the predictors of poor outcomes in these patients .

Episodes were defined on the basis of a Glasgow Coma Score (GCS) of less than 12 for more than six hours . Many acutely ill children are not fully conscious because pathologic processes may affect the parts of the central nervous system that mediate consciousness; alteration in the state of consciousness is a common feature of many different conditions.

Many of these children make a full neurological recovery. However, depending on the underlying etiology non-traumatic coma may cause considerable mortality and morbidity in pediatric age group .

ELIGIBILITY:
Inclusion Criteria:

* disturbed conscious level
* Children's family signed consent of approval to participate in the study

Exclusion Criteria:

1. Children aged <2 months or >18 years.
2. Coma of traumatic etiology.
3. Coma as part of an anticipated terminal illness.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted in Assiut University Hospital with impaired consciousness .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of recovery from coma | 1 month
  clinical evaluation of the recovery symptoms and signs

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Zaka, Principal Investigator — World Health Organization